

# Information notice

Non-comparative phase II pilot trial to evaluate the ability of a combination of raltegravir + etravirine to maintain virological success in HIV-1-infected patients of at least 45 years of age with a plasma viral load of less than 50 copies/mL on antiretroviral therapy including a boosted protease inhibitor.

Version 2.0, dated 03/18/2015, approved by the CPP on 05/15/2015

# **Coordinating Investigator:**

Prof. Christine Katlama, Pitié-Salpêtrière Hospital, Paris.

#### **Scientific Director:**

Prof. Jacques Reynes, Montpellier University Hospital.

#### **Trial Sponsor:**

National Institute of Health and Medical Research - National Agency for Research on AIDS and Viral Hepatitis (Inserm - ANRS) 101 rue de Tolbiac, Paris 75013.

- This notice is designed to help you decide whether or not to participate in the trial described below.
- You are free to answer yes or no to the question asked: do you want to participate in the trial?
- You have the right to take as much time as you need to think about it, to discuss this trial and to ask anyone you want whatever you want to know about it.
- If you do not wish to participate, you will still continue to receive the best possible care
- You can change your mind at any time and ask to withdraw from the trial. You will continue to benefit
  from the best care that your doctor can offer you. We ask only that you inform your doctor of your
  decision as soon as possible.

Page 1 of 11

The words underlined in the text are explained in the glossary.

# **Glossary**

**Biobank:** A bank of biological samples kept for research purposes.

Data: Information collected as part of the trial.

Right of access: The right to see the data concerning you.

**Anonymized data**: Your name and surname are removed from all medical records and replaced with a code. Only the doctor and people with a right of access to the medical data are aware of the link between your identity and this code.

**Right of opposition**: The right to oppose the transmission of your data by the investigating doctor to the sponsor. The exercise of this right terminates your participation in the trial.

Right of rectification: The right to request that the correction of your data in the event of an error.

**Samples**: Samples taken from people participating in the trial (e.g. blood, cells, etc.). In general, the samples are stored in a **Biobank** centralized at the ANRS.

**Consent form**: A document in which you declare that you have read the terms of participation in the trial and give your consent to participate.

**Coordinating investigator**: The doctor supervising the running of the trial at the various participating centers.

**Investigating doctor of the trial (or investigator)**: The doctor following you in the framework of the trial. He/she may be your regular doctor, or another doctor involved in the trial.

**Bone densitometry**: A painless radiological examination measuring the mineral content of the bone, and the percentage of fat and lean mass in the limbs and trunk.

Pre-inclusion: The time point at which all conditions are met for your participation in the trial.

**Sponsor**: The organization legally and financially responsible for the trial.

**Substudy**: A study carried out only on some of the people participating in the trial.

Adipose tissue: A tissue that contains fat.

**Integrase inhibitor:** A molecule that blocks a viral enzyme, integrase, which allows the virus to enter the cell's nucleus to multiply.

**Non-nucleoside reverse transcriptase inhibitor:** A molecule that blocks a viral enzyme, reverse transcriptase, the role of which is to convert the viral genome into DNA that can integrate into the genome of the host cell.

# In this notice you will find:

1. The objectives of the trial

4

2. The conditions for participation in the trial


3. A schema for the trial


4. The trial treatments

5

| 5. Sexuality, contraception, and pregnancy | 6 |
|---|---|
| 6. What are the constraints linked to participation in this trial? | 6 |
| 7. The progress and timetable of the trial | |
| 8. Expected benefits and possible risks | g |
| 9. Monitoring | |
| 10. Alternatives | g |
| 11. What will happen at the end of the trial | g |
| 12. What are your rights? | g |
| 13. Information about the fate of your samples at the end of the trial | 11 |

You will find a <u>consent form</u> on the last page: this signed document attests to your willingness to participate in the trial and contains the contact details of the <u>investigating doctor</u> of the trial, whom you can contact if necessary.

To whom it may concern,

The investigating doctor of the ANRS 163 ETRAL trial would like to invite you to participate in this trial.

You have been on antiretroviral therapy including at least one boosted protease inhibition for the treatment of HIV infection for at least six months. This treatment makes it possible to control your viral load, that is, it prevents the multiplication of the virus in the blood (resulting in what we call an "undetectable plasma viral load"). This treatment also increases the number of CD4 cells in the blood, improves survival, and slows disease progression.

Despite the considerable clinical progress achieved in patients whose virus is under control, vascular (angina pectoris or myocardial infarction), lipid (increases in cholesterol and triglyceride levels), renal (a decrease in the filtration rate of the kidney), or bone (decrease in bone density) complications may emerge over time. They are related to the persistent inflammation due to HIV, and to certain molecules used in antiretroviral treatments, such as, nucleoside or nucleotide analogs (tenofovir (Viréad®, Truvada®) or abacavir (Ziagen®, Kivexa®)) and protease inhibitors (atazanavir (Réyataz®), darunavir (Prézista®) lopinavir / r (Kalétra®)). The frequency of these events also increases with age and increasing patient life expectancy. Today, almost 40% of patients treated in French hospitals at least 50 years old. A comparison between HIV-positive and HIV-negative patients has shown that the frequency of complications is higher in HIV-positive patients and that these complications occur earlier.

Some of the most recent classes of antiretroviral therapy or drugs are both effective against HIV and have little effect on lipid balance, bones, or <u>adipose tissue</u>.

We are inviting you to participate in a trial evaluating a new strategy combining two powerful antiretroviral drugs that are well known and have been marketed for several years:

- Raltegravir (or Isentress®), which has been available since 2008, belongs to the new class of <u>integrase inhibitors</u> (integrase allows the virus to enter the nucleus of the cell to multiply).
- Etravirine (or Intelence®), which belongs to the second generation of <u>non-nucleoside reverse transcriptase</u> <u>inhibitors</u>, blocks a viral enzyme, reverse transcriptase, which converts the viral genome into DNA capable of integrating into the genome of the host cell (see the *Trial treatments* section).

# 1. Objectives of the trial

The objective of the trial is to determine whether this new combination of two antiretroviral molecules — raltegravir (Isentress®) and etravirine (Intelence®) — makes it possible to maintain an undetectable HIV viral load while reducing potential side effects, such as cardiovascular, bone, kidney, or adipose tissue distribution disorders.

This trial includes two substudies to evaluate the following parameters:

- The DXA substudy: changes in the distribution of <u>adipose tissue</u> in the body and in bone mineral density. This substudy will involve a painless radiological examination for measuring the mineral content of the bone, and the percentage of fat and lean mass in the limbs and trunk, which will be performed at regular intervals (day (D) 0, week (W) 48, W96) for 80 participants.
- The semen substudy: measurements of HIV RNA viral load and the residual concentrations of raltegravir (Isentress®) and etravirine (Intelence®) in a sample of sperm fluid collected at W48 from 20 male participants.

# 2. The conditions for participation in the trial

If you decide to participate in this trial, a first visit, the "pre-inclusion visit", will take place 2 to 4 weeks before the start of the trial. During this visit, the doctor will assess your state of health: clinical examination, weight, height; blood and urine samples will also be collected. Your doctor will ask you about your medical history, to check that you are eligible to participate in the trial.

## The principal conditions for participation in this trial are as follows. You must:

- Be at least 45 years old
- Be infected with HIV-1
- Have been on stable antiretroviral treatment for at least six months
- Have a CD4 lymphocyte count above 200/mm<sup>3</sup>
- Have had an undetectable viral load (i.e. less than 50 copies/mL) for at least 24 months
- Have never been treated with raltegravir (Isentress®) and etravirine (Intelence®)
- -Not take prohibited drugs during the trial (see the list in the *Trial treatments* section)
- Accept the constraints imposed by the trial (see the paragraph *What are the constraints linked to participation in the trial?* section)
- Be affiliated to or be a beneficiary of a social security regime (State Medical Aid or AME is not a social security regime)
- Have signed the <u>consent form</u>: this form must be signed before any examination (e.g. blood test, scan, etc.) is carried out as part of the trial
- Not participate in another trial at the same time as this one

#### The following situations are incompatible with participation in the trial:

- Being pregnant or breastfeeding
- Having chronic hepatitis B or C (treated during the 24 months of the trial)
- Anti-hypercholesterolemia and/or anti-diabetic treatment initiated in the 3 months preceding your participation in the trial

If, after checking these conditions, the investigator decides that you cannot participate in this trial, he/she will decide, with you, which treatment is best suited to your situation.

# 3. Schema for the trial

Once the eligibility criteria have been verified, you can start the trial.

All participants will replace their usual antiretroviral therapy with raltegravir (Isentress®) plus etravirine (Intelence®).

Therefore, all trial participants will receive the same treatment: raltegravir (Isentress®) and etravirine (Intelence®).

The duration of participation in the trial is 96 weeks (approximately two years).

The maximum total duration of the trial is estimated at four years, including the time required to include all the trial participants.

We to include 160 participants from several hospitals in France and Spain.

# 4. Trial treatments

# Raltegravir (Isentress®): what you should know

Raltegravir (Isentress®), developed by the Merck Sharp & Dohme Ltd laboratory, has been marketed in France since January 2008.

Raltegravir (Isentress®) blocks the action of an enzyme (protein) called "integrase". It is produced in the form of tablets and must be taken at a dose of 1 tablet twice daily (i.e. 2 tablets per day).

The tolerance of raltegravir (Isentress®) is generally good. However, like most treatments, it can cause certain adverse effects, the main ones being:

- Diarrhea, nausea (feeling sick) and headache (may affect more than 1 in 10 people)
- Insomnia (difficulty sleeping), dizziness, bloating, stomachache, flatulence (gas), vomiting, rash, weakness, fatigue (may affect 1 to 10 users in 100)
- Contact your doctor immediately if you develop a cutaneous (skin) reaction. Skin reactions and life-threatening severe allergic reactions have been reported in some people receiving this medicine.
- Inform your doctor if you have a history of depression or psychiatric illness. Depression, including suicidal thoughts and behavior, has been reported in some people taking this medication, especially those with a history of depression or psychiatric illness.

# Etravirine (Intelence®): what you should know

Etravirine (Intelence<sup>®</sup>), developed by Janssen Cilag Laboratories, has been marketed in France since August 2008.

It is produced in the form of tablets and must be taken at a dose of 1 tablet twice daily (i.e. 2 tablets per day).

Etravirine is a <u>non-nucleotide reverse transcriptase inhibitor</u>.

Tolerance to etravirine is generally good, but like most treatments, it can have certain adverse effects, the main ones being:

- Skin rashes that are usually mild to moderate. However, a very serious and potentially life-threatening rash has been reported in rare cases. It is therefore important that you contact your doctor immediately if you develop a rash.
- Nausea, stomach problems (diarrhea, stomachache, indigestion), headache, dizziness, tiredness (may affect less than 1 in 10 people).

- Risk of myocardial infarction (frequency: less than 1 in 10 people).

## Doses of raltegravir (Isentress®) and etravirine (Intelence®):

The table below specifies the dose and number of doses of the treatments that you will take as part of this trial:

| Who? | Medicine | Form | Morning | Evening | How to take it |
|---|---|---|---|---|---|
| | Raltegravir 400 mg (Isentress®), | Pink oval tablets | 1 | 1 | After a meal |
| All participants | Etravirine 200 mg (Intelence®), | White oval tablets | 1 | 1 | After a meal |

If you want more information about these treatments, do not hesitate to talk to your doctor.

## Tell your doctor before taking other medicines during the trial:

It is important to tell your doctor about the medicines that you take or wish to take (with or without a prescription) during the trial.

The following drugs are **formally contraindicated** and must not be taken in combination with the trial treatments because they may interact with or limit the efficacy of the anti-HIV treatments:

- Antiplatelet agents: Clopidogrel (Plavix®), prasugrel (Effient®), ticagrelor (Brilique®), ticlopidine (Ticlid®), flurbiprofene (Antadys® Cebutid®).
- Anti-infection agents: Rifampicine (Rifampicine® Rifadin® RofactMC Rifater®), rifapentine (Priftin®).
- · Certain herbal medicines containing St. John's Wort.
- Anti-epileptic agents: Carbamazepine (Tegretol®), phenobarbital, phenytoine (Dilantin®).
- Other drugs: Avanafil (Stendra™), triazolam (Halcion®).

If you have any questions about these medicines, do not hesitate to talk to your doctor.

# 5. Sexuality, contraception, and pregnancy

It is very important to use a condom during sex, because treatment for HIV does not always prevent the transmission of HIV and other sexually transmitted infections.

Raltegravir (Isentress®) and etravirine (Intelence®) have not been evaluated in pregnant women. Their effects on the unborn child are not known. It is therefore important not to take any risks and not to become pregnant during the trial. You should discuss the contraceptive method best suited to your situation with your doctor. If you, nevertheless, discover that you are pregnant during the trial, you should immediately tell your doctor.

# 6. What are the constraints linked to participation in the trial?

During this trial, medical examinations will be slightly more frequent than during your usual follow-up. You should expect:

- A <u>pre-inclusion</u> visit and 10 follow-up visits during the two years of participation.
- Blood tests at each visit and questionnaires to be completed at certain visits.

If you agree to take part in one or both of the two proposed <u>substudies</u>, you must also be available for the examinations or blood tests for these <u>substudies</u>: <u>bone densitometry</u> (a painless radiological examination that measures the mineral content of bone and the percentages of fat and lean mass in the limbs and trunk) and sperm collection.

For your safety and for the success of the trial, it is important to follow the visit schedule as closely as possible. Given the importance of keeping to the timetable for the trial, the medical team in charge of your follow-up in the trial will do their utmost to facilitate this. You will be in contact with the clinical research team of your center, who will give you your schedule and all the telephone numbers that might prove useful for the smooth running of your participation. If you cannot come for a consultation or provide a sample, remember to tell your doctor.

Your agreement to participate in this trial implies that you accept the constraints imposed by the scheduled examinations.

Do not hesitate to ask the <u>investigating doctor</u> all the necessary questions on this subject. If you wish, he/she can give you information about your follow-up in the trial at each consultation.

# 7. The progress and timetable of the trial

If you agree to participate in the trial, you will sign a <u>consent form</u> before the first examination related to the trial. You will have a total of 11 visits spread over the two years of your participation in the trial:

"Pre-inclusion" visit: the <u>investigating doctor</u> will ask you about your medical history and perform a clinical examination and blood tests to make sure that you can participate in the trial.

If all the conditions for participation are met:

Visit D0: corresponds to the first dose of raltegravir (Isentress®) and etravirine (Intelence®). This visit takes place 2 to 4 weeks after the pre-inclusion visit.

There will be 9 other visits: W2, W4, W12, W24, W36, W48, W64, W80, and W96 (see the trial calendar).

During these visits, the <u>investigating doctor</u> will take blood samples for routine blood tests, such as blood sugar, the measurement of viral load (measurement of the amount of virus in the blood), or counts of CD4 lymphocytes. Other blood samples will be used to carry out more specific blood tests, such as determinations of the amount of the trial drugs in your blood.

Some samples/blood samples will be analyzed immediately, and others will be kept for analysis at the end of the trial.

You will be asked for a urine sample at visits W-6/W-4, W4, W12, W24, W48, W80, and W96, to check for protein or glucose (sugar) in your urine, these substances normally being present in only very small amounts.

Blood <u>samples</u> for storage will be sent to the French Blood Establishment (EFS) in Beynost (France) to constitute a <u>biobank</u>. Each <u>sample</u> will be labeled and numbered anonymously (your name will not be indicated).

The samples from the <u>biobank</u> can be used for additional studies. If these additional studies involve genetic testing, you will be asked for consent for such testing.

You can specify in your <u>consent</u> that you do not wish your samples to be kept in the <u>biobank</u> for use in future research.

#### **Substudies**

If you are volunteering for the DXA substudy, to evaluate changes in the distribution of fat in your body and changes in bone mineral density, bone densitometry will be performed on D0 and at W48 and W96 (80 participants).

Patients wishing to participate in the semen substudy, which aims to measure the viral load of HIV and the residual concentration of raltegravir (Isentress®) and etravirine (Intelence®) in sperm fluid, will provide a sperm sample at W48 (20 participants).

# The questionnaires and self-administered questionnaires to be completed during the trial

- "Quality of life" and "compliance" self-administered questionnaires: These are anonymized questionnaires, on paper, that you will complete on your own. At no time will we be able to intervene your responses. The self-administered "compliance" questionnaire will tell us whether you are taking your treatments as prescribed by your doctor. If this is not the case, your doctor will try to understand why and work with you to try to find a solution.

## **Trial Calendar**

| | Pre-<br>inclusion*<br>(W-6/W-4<br>to<br>W-2) | D:<br>Start of<br>treatment | W2 | W4 | W12 | W24 | W36 | W48 | W64 | W80 | W96 | In case of virological failure |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Signature of consent form | | | | | | | | | | | | |
| Clinical examination | | | | | | | | | | | | |
| Quality of life self-<br>administered<br>questionnaires | | | | | | | | | | | | |
| Compliance questionnaire | | | | | | | | | | | | |
| Come to the consultation after a period of at least 12 h without eating | | | | | | | | | | | | |
| Pregnancy test (1) | | | | | | | | | | | | |
| Urine sample | | | | | | | | | | | | |
| DXA / Bone densitometry (substudy) | | | | | | | | | | | | |
| Sperm sample<br>(substudy) | | | | | | | | | | | | |
| Amount of blood for the ETRAL trial (without storage in the biobank) | 29 mL (7 tubes) | 22 mL<br>(6 tubes) | 0 mL | 19 mL<br>(5<br>tubes) | 22 mL<br>(6<br>tubes) | 25 mL<br>(7<br>tubes) | 7 mL<br>(1<br>tubes) | 25mL<br>(7<br>tubes) | 7 mL<br>(1<br>tubes) | 16 mL<br>(4<br>tubes) | 25 mL<br>(7<br>tubes) | 14 mL<br>(2 tubes) |
| Additional blood for the biobank | 0 mL | 45 mL<br>(7 tubes) | 21 mL<br>(3<br>tubes) | 21 mL<br>(3<br>tubes) | 21 mL<br>(3<br>tubes) | 21 mL<br>(3<br>tubes) | 21 mL<br>(3<br>tubes) | 45 mL<br>(7<br>tubes) | 21 mL<br>(3<br>tubes) | 21 mL<br>(3<br>tubes) | 45 mL<br>(7<br>tubes) | 7 mL (1<br>tubes) |
| Total amount of blood collected (mL) | 29 mL (7<br>tubes) | 67 mL<br>(13 tubes) | 21 mL<br>(3<br>tubes) | 40 mL<br>(8<br>tubes) | 43 mL<br>(9<br>tubes) | 46 mL<br>(10<br>tubes) | 28 mL<br>(4<br>tubes) | 70 mL<br>(14<br>tubes) | 28 mL<br>(4<br>tubes) | 37 mL<br>(7<br>tubes) | 70 mL<br>(14<br>tubes) | 21 mL (3 tubes) |

\*Pre-inclusion: takes place 2 to 4 weeks before the start of treatment. W: week

<sup>(1)</sup> The pregnancy test is carried out only for women of childbearing age at W-6/W-4 and then at subsequent visits if pregnancy is suspected.

# 8. Expected benefits and possible risks

#### **Expected benefits**

- The antiretroviral drugs that you will receive as part of the ANRS 163 ETRAL trial have shown, separately, to have virological efficacy, with raltegravir (Isentress®) having a lesser effect on lipid profile and bones.

You will benefit from participation if the trial shows that the raltegravir (Isentress®) + etravirine (Intelence®) combination controls viral replication, is well tolerated, and reduces the frequency of complications associated with HIV infection and your previous treatment.

- You will benefit from more frequent monitoring and more detailed examinations.
- You will be involved in research, the results of which may be of benefit to other people.

#### Possible risks

- Raltegravir (Isentress®) and etravirine (Intelence®) can cause known (as described in the *Trial treatments* section) or unknown adverse effects.
- The trial treatment should control viral replication and ireduce the complications of HIV infection and your previous treatment. However, there is a risk of replication. You will be monitored closely to detect any rise in HIV viral load.
- Blood tests may cause bruising at site of puncture, on the day of the examination and on the following two to three days.

# 9. Monitoring

During the trial if, for example, your health deteriorates and other treatments are preferable, or if justified by adverse effects, you can decide, with your doctor, to stop the trial treatment at any time, while continuing your monitoring.

Throughout the trial, scientific committees will monitor the study for adverse effects or failures of raltegravir (Isentress®) and etravirine (Intelence®). These committees ensure the safety of those involved in the trial and oversee the running of the trial. If necessary, for safety reasons, for example, they can decide to end the trial or to modify the way in which it is performed.

# 10. Alternatives

You should know that your participation in the trial is free and voluntary. You can decide to refuse to participate in the trial and remain on your current treatment. Your decision to agree or refuse to participate in this trial will not change the quality of your medical care.

# 11. What will happen at the end of the trial?

Raltegravir (Isentress®) and etravirine (Intelence®) are already sold in France. If the final results of the trial are conclusive, your doctor may wish to consider continuing with this combination. At the end of the trial, participants will be able to discuss their results and their experience of participation in the trial.

The overall results of the trial will be communicated to the participants after the trial has ended.

# 12. What are your rights?

#### Do not forget that you can:

- Take as long as you need to think before deciding to participate in this trial
- Leave the trial at any time, without giving a reason, by simply telling your doctor
- Find out about your health
- Be informed of any serious events occurring during the trial
- Be informed of your results and of the overall results of the trial
- Check and correct data concerning you
- Oppose the transmission of data concerning you
- Obtain compensation in the event of harm

#### Your data:

As part of the trial in which you are being asked to participate by the National Agency for Research on AIDS and Viral Hepatitis (ANRS), your personal <u>data</u> will be processed as part of the analysis of the results of the trial with respect to its objectives, which have been presented to you.

To this end, the medical <u>data</u> concerning you and the <u>data</u> relating to your lifestyle, and, insofar as these <u>data</u> are necessary for the trial, your ethnic origins, and sex life, will be transmitted to the <u>sponsor</u> of the trial or to individuals or companies acting on the sponsor's behalf, in France or abroad.

These <u>data</u> will be identified by a code number. These <u>data</u> may also be transmitted to French or foreign health authorities (Medicines Agency, etc.) or to other ANRS partners, under conditions of confidentiality.

In accordance with the provisions of the law relating to data processing and freedoms, you have the <u>right of access</u> and <u>rectification</u>. You also have the <u>right to oppose</u> the transmission of <u>data</u> covered by professional secrecy that may be used in the context of this trial and be processed. The exercise of this right will terminate your participation in the trial.

You can also access all of your medical <u>data</u> directly or through a doctor of your choice, in accordance with the provisions of article L 1111-7 of the French Public Health Code.

If you have any questions about these rights, you can contact the doctor following you during the trial. If desired, information about the trial and your participation will be shared with your general practitioner.

This trial received was approved by the Personal Protection Committee (CPP) on 04/16/2014 and authorized by the ANSM on 04/04/2014.

The sponsor of this trial, Inserm-ANRS, has taken out civil liability insurance in the event of harm, in accordance with the provisions of the French Public Health Code, with HDI Gerling (Tours opus 12, 77 Esplanade de la Défense 92914 PARIS LA DEFENSE).

The French Public Health Code also guarantees compensation to anyone suffering harm due to participation in research.

| <b>ANRS</b> | 163 | ETR | AL | Trial |
|-------------|-----|-----|----|-------|
|-------------|-----|-----|----|-------|

To whom it may concern,

As specified in the information notice specific to the ANRS 163 ETRAL trial, in which you are invited to participate, blood samples, urine samples, and (possibly) a semen sample will be taken.

If the blood and semen <u>samples</u> are not completely used up at the end of this trial, they may be used for scientific research on HIV unless you object.

The remaining <u>samples</u>:

- Will be stored at the EFS (French Blood Establishment Beynost site), under the control of its logistics management, on behalf of the ANRS, and under the scientific responsibility of the common service 10-US019 of Inserm (Paul Brousse Hospital, Villejuif)
- May be supplied free of charge, and under certain conditions, to other national or international private or public research groups, under conditions guaranteeing the confidentiality of your <u>data</u>
- May not, in any case, be used for the examination of genetic characteristics without new written consent from you.

# You may freely, and at any time, object to this further use for research purposes, by contacting the <u>investigating doctor of the trial</u>.

Your decision will have no consequences for your participation in the ANRS 163 ETRAL trial or your medical care.

| Name, address, and contact details. |
|-------------------------------------|

In accordance with the law, no remuneration can be paid to you.

The transferred <u>samples</u> cannot be sold.

For <u>sample</u> management, the EFS uses a computer file authorized by the French National Commission for Data Protection (CNIL). This file contains <u>anonymized data</u> for the identification of <u>samples</u>.

| ANRS 163 | BETRAL T | rial | ( | Consent Form |
|----------|-----------|-------------|-------------|--------------|
| Country | Center No | Patient No. | Letter code | 4 |

| Version 2.0 of 03/18/2015, approved by the CPP on 05/15/2015 Sponsor: Inserm-ANRS Coordinating investigator: Prof. Christine Katlama Ms, Mr |
|---|
| I certify: having received information notice version 2.0 dated 03/18/2015, that I have had the opportunity to ask all the questions I wished on the nature, objectives, potential risks, and constraints relating to my participation in this trial, and that I have had sufficient time to reflect between receiving this information and giving my consent. I understand the constraints (more frequent visits, numerous blood samples) and the benefits linked to my participation in this trial, which will last approximately 2 years. |
| I understand that I am free to discontinue my participation in this trial at any time, without having to explain why, but I will do my best to inform the doctor. This will not affect the quality of my subsequent care. |
| I have been reassured that the decisions that are necessary for my health will be made at all times, in accordance with the state of knowledge on HIV. |
| I have noted that blood samples and a semen sample (if I participate in the semen substudy) will be taken during the trial and stored anonymously. They will make it possible to carry out the planned analyses for this trial. |
| I accept that the data recorded during this trial will be collected, processed, and computerized. I understand that the right of access laid down in the modified law of January 6, 1978 relating to data processing, files, and freedoms, can be exercised at any time, through the doctor following me in the trial, and that I can exercise my right of rectification and opposition. |
| I accept that the scientists involved in this trial, and the individuals authorized by the health authorities in France and abroad, may have access to the information, under strict conditions of confidentiality. |
| My consent in no way relieves the organizers of the trial of their responsibilities. I retain all my statutory rights. |
| At the end of the trial, I may be informed of the overall results through the investigating doctor of the trial. |
| I have been informed by the explanatory notice that my blood and/or semen samples may be used at the end of the trial for other research on HIV infection, <b>unless I oppose this</b> . |
| I authorize the storage of my blood samples for future research. I oppose the storage of my blood samples for future research. They will be destroyed at the end of the trial. |
| I agree to participate in the DXA substudy "Distribution of fat mass and bone mineral density" |
| I agree to participate in the seminal sub-study "Measurement of RNA-HIV viral load in semen" |
| I authorize the storage of my sperm samples for further research. |
| I freely agree to participate in this test under the conditions specified in the information notice Participant's signature |
| Date |
| I, the undersigned, Dr/Pr certify that I have communicated to the participant all the useful information relating to this trial, that I have answered his questions and obtained his consent. Date |

| ANRS 163 ETRAL Trial | <b>Consent Form</b> | |
|---|---|---|
| Country Center No. Patient No. | Letter code | |
| Write or place a label Name of the unit: Address: Telephone: | | Doctor's signature |
| INVESTIGATOR CORV. ( | ' | |

INVESTIGATOR COPY (a copy is made for the sponsor)

## Version 2.0 dated 03/18/2015, approved by the CPP on 05/15/2015

Sponsor: Inserm-ANRS Coordinating investigator: Prof. Christine Katlama

Ms, Mr (first last name)
I certify:



and

having received information notice version 2.0 dated 03/18/2015, that I have had the opportunity to ask all the questions I wished on the nature, objectives, potential risks, and constraints relating to my participation in this trial, and that I have had sufficient time to reflect between receiving this information and giving my consent.

I understand the constraints (more frequent visits, numerous blood samples) and the benefits linked to my participation in this trial, which will last approximately 2 years.

I understand that I am free to discontinue my participation in this trial at any time, without having to explain why, but I will do my best to inform the doctor. This will not affect the quality of my subsequent care.

I have been reassured that the decisions that are necessary for my health will be made at all times, in accordance with the state of knowledge on HIV.

I have noted that blood samples and a semen sample (if I participate in the semen substudy) will be taken during the trial and stored anonymously. They will make it possible to carry out the planned analyses for this trial.

I accept that the data recorded during this trial will be collected, processed, and computerized. I understand that the right of access laid down in the modified law of January 6, 1978 relating to data processing, files, and freedoms, can be exercised at any time, through the doctor following me in the trial, and that I can exercise my right of rectification and opposition.

I accept that the scientists involved in this trial, and the individuals authorized by the health authorities in France and abroad, may have access to the information, under strict conditions of confidentiality.

My consent in no way relieves the organizers of the trial of their responsibilities. I retain all my statutory rights.

At the end of the trial, I may be informed of the overall results through the investigating doctor of the trial.

I have been informed by the explanatory notice that my blood and/or semen samples may be used at the end of the trial for other research on HIV infection, **unless I oppose this**.

| I authorize the storage of my blood samples for future research. | I oppose the storage of my blood samples for future research. They will be destroyed at the end of the trial. |
|---|---|
| I agree to participate in the DXA substudy "Distribution of fat mass and bone mineral density" | |
| I agree to participate in the seminal sub-study "M | Measurement of RNA-HIV viral load in semen" |
| I authorize the storage of my sperm samples for further research. | I oppose the storage of my sperm samples for future research. They will be destroyed at the end of the trial. |

| I freely agree to participate in this trial under the conditions | |
|---|---|
| specified in the information notice | Participant's signature |
| Date L | |

| ANRS 163 ETRAL Trial Consent Form | |
|---|---|
| Country Center No. Patient No. Letter code | |
| I, the undersigned, Dr/Pr certify that I have communicated to the participant all the useful informations/her questions and obtained his/her consent. Date | tion relating to this trial, that I have answered |
| Write or place a label Name of the unit: | Doctor's signature |
| Address: | |
| Telephone: | |

**CMG Inserm UMR S 1136 COPY** 

| ANRS 16 | 3 ETRAL T | rial | ( | Consent Form |
|-----------|---------------|-------------|-------------|--------------|
| ا لـــــا | ا لــلـــلـــ | | | |
| Country | Center No | Patient No. | Letter code | <b>.</b> |

**Sponsor: Inserm-ANRS** 

I freely agree to participate in this trial under the conditions

specified in the information notice

Date LL LL

## Version 2.0 dated 03/18/2015, approved by the CPP on 05/15/2015

| | • | 0 | 8 | |
|--------|---|---|---|-----------------------|
| Ms, Mr | | | | (first and last name) |

Coordinating investigator: Prof. Christine Katlama

## I certify:

having received information notice version 2.0 dated 03/18/2015, that I have had the opportunity to ask all the questions I wished on the nature, objectives, potential risks, and constraints relating to my participation in this trial, and that I have had sufficient time to reflect between receiving this information and giving my consent.

I understand the constraints (more frequent visits, numerous blood samples) and the benefits linked to my participation in this trial, which will last approximately 2 years.

I understand that I am free to discontinue my participation in this trial at any time, without having to explain why, but I will do my best to inform the doctor. This will not affect the quality of my subsequent care.

I have been reassured that the decisions that are necessary for my health will be made at all times, in accordance with the state of knowledge on HIV.

I have noted that blood samples and a semen sample (if I participate in the semen substudy) will be taken during the trial and stored anonymously. They will make it possible to carry out the planned analyses for this trial.

I accept that the data recorded during this trial will be collected, processed, and computerized. I understand that the right of access laid down in the modified law of January 6, 1978 relating to data processing, files, and freedoms, can be exercised at any time, through the doctor following me in the trial, and that I can exercise my right of rectification and opposition.

I accept that the scientists involved in this trial, and the individuals authorized by the health authorities in France and abroad, may have access to the information, under strict conditions of confidentiality.

My consent in no way relieves the organizers of the trial of their responsibilities. I retain all my statutory rights.

At the end of the trial, I may be informed of the overall results through the investigating doctor of the trial.

I have been informed by the explanatory notice that my blood and/or semen samples may be used at the end of the trial for other research on HIV infection, **unless I oppose this**.

| future research.<br>hey will be destroyed at the end of the trial. |
|---|
| I agree to participate in the DXA substudy "Distribution of fat mass and bone mineral density" |
| I agree to participate in the semen substudy "Measurement of HIV-RNA viral load in semen" |
| I oppose the storage of my sperm samples for future research. hey will be destroyed at the end of the trial. |
| t |

Participant's signature

| ANRS 163 ETRAL Trial Consent Form | |
|--------------------------------------------|--------------------|
| Country Center No. Patient No. Letter code | |
| I, the undersigned, Dr/Prof | |
| Date | |
| Write or place a label Name of the unit: | Doctor's signature |
| Address: | |
| Telephone: | |

PATIENT'S COPY (attached to the notice)